CLINICAL TRIAL: NCT04210791
Title: Autologous Stem Cell Transplantation for Patients With AL Amyloidosis
Status: Enrolling by invitation | Type: Observational
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhi-Hong Liu, MD, Professor, Nanjing University School of Medicine
Other Study IDs: NJCT-1901
Record Dates: First submitted 2019-12-14; First posted 2019-12-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: AL Amyloidosis; Plasma Cell Dyscrasia
Keywords: AL amyloidosis; autologous stem cell transplantation; induction therapy; bortezomib; lenalidomide; ixazomib; daratumumab; melphalan
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Paraproteinemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study mainly evaluated the efficacy and safety of autologous stem cell transplantation for the treatment of AL amyloidosis, the role of induction and maintenance therapy in autologous stem cell transplantation, and the long-term efficacy and prognosis risk factors of autologous stem cell transplantation for the treatment of AL amyloidosis.

DETAILED DESCRIPTION:
This study is divided into two parts. In the first part, the investigators retrospectively analyze the data of patients with AL amyloidosis who treated with autologous stem cell transplantation from July 2010 to December 2019. All patients had a biopsy-proven disease by positive Congo red stain with a concomitant demonstration of plasma cell dyscrasia. Organ involvement was established according to the criteria established at the 10th International Symposium on Amyloid and Amyloidosis. The protocol of ASCT included mobilization with colony-stimulating factor alone and conditioning with high-dose melphalan 140 or 200 mg/m2. In addition to analyzing the efficacy and safety of all the patients, the investigators also analyzed the difference in efficacy between patients in different subgroups. For example, subgroups divided according to different induction treatment regimens; subgroups divided according to different plasma cell FISH data and FCM data; subgroups divided according to the degree of organ involvement, and subgroups divided according to different maintenance treatment regimens.

In the second part of the study, the investigators will conduct a prospective study to explore the best autologous stem cell transplantation treatment protocol for AL amyloidosis. The protocol includes the induction therapy with bortezomib and daratumumab before ASCT, the maintenance treatment with lenalidomide after ASCT, and the treatment options for recurrence after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* aged 18-75 years;
* Patients with newly diagnosed AL;
* Appropriate for autologous hematopoietic stem cell transplantation;
* Abnormal M protein or free light chain detected in serum and/or urine
* ECOG score 0-2 points;
* Subjects (or their legal representatives) must sign an informed consent document indicating understanding the purpose of and procedures required for the study and willingness to participate in the study.

Exclusion Criteria:

* Pregnant and breastfeeding women;
* Subjects suffering from multiple myeloma;
* hypersensitivity to any treatment drugs;
* Subjects have severe cardiovascular disease;
* Subjects have a serious physical disease and mental illnesses;
* Other conditions that researchers consider are not suitable for transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients had an amyloid disease, which was confirmed by biopsy and documented plasma cell dyscrasia; the AL amyloidosis diagnosis and the assessment of organ involvement were based on previous consensus criteria. All patients had received autologous stem cell transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years
  the 5 years overall survival after autologous stem cell transplantation.
progression-free survival | 5 years
  the 5 years progression-free survival after autologous stem cell transplantation.
hematological complete response rate | 1 year
  the 1 year hematologic complete response rate after autologous stem cell transplantation.
organ response rate | 1 year
  the 1 years organ response rate after autologous stem cell transplantation.

SECONDARY OUTCOMES:
hematological overall response rate | 1 year
  the 1 years hematologic overall response rate after autologous stem cell transplantation.
the relapse rate of complete remission participants | 5 years
  the relapse rate of complete remission participants after autologous stem cell transplantation.
the rate of Minimal Residual Disease-negative participants | 5 years
  the rate of Minimal Residual Disease-negative participants after autologous stem cell transplantation.
the median time form stem cell transplantation to next treatment | 5 years
  the median time form stem cell transplantation to next chemotherapy or antibody treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, MD, Study Director — Nanjing University School of Medicine
Locations (1):
- National Clinical Research Center of Kidney Diseases, Jinling Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Zhang Y, Guo J, Chen W, Zhao L, Huang X. Risk factors, treatments and outcomes of patients with light chain amyloidosis who relapse after autologous stem cell transplantation. Bone Marrow Transplant. 2024 Mar;59(3):350-358. doi: 10.1038/s41409-023-02185-z. Epub 2023 Dec 26. PMID 38148411